CLINICAL TRIAL: NCT01449240
Title: A Cerebrospinal Fluid Collection Study in Pediatric and Adult Patients With Hunter Syndrome
Brief Title: Collection and Study of Cerebrospinal Fluid in Patients With Hunter Syndrome
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: HGT-HIT-072
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Results first posted 2014-12-05 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Hunter Syndrome
Keywords: Hunter syndrome; Mucopolysaccharidosis II; Iduronate 2-Sulfatase Deficiency; Lumbar puncture; Cerebrospinal fluid (CSF); Pediatric; Adult; Biomarkers
MeSH Terms: conditions — Mucopolysaccharidosis II

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CSF and urine samples will be retained and analyzed for glycosaminoglycans (GAGs), including sulfated DS/HS oligosaccharides, GAG-degradation products, and other biomarkers of CNS or lysosomal function.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Approximately 5 adults (equal to or not less than 18yrs old) and 5 children (equal to or not over 18yrs old)
  Interventions: Other: No treatment

INTERVENTIONS:
Other: No treatment

SUMMARY:
The purpose of the study is to collect data on CSF biomarkers in patients with Hunter Syndrome that would serve as reference data for comparison with cognitively impaired patients with Hunter syndrome, patients with other lysosomal storage diseases, or other diseases with CNS involvement.

DETAILED DESCRIPTION:
To determine levels of glycosaminoglycans (GAGs), including dermatan sulfate (DS) and heparan sulfate (HS), GAG-degradation products, and other biomarkers of central nervous system (CNS) and lysosomal function in cerebrospinal fluid (CSF) in pediatric and adult patients with Hunter syndrome.

ELIGIBILITY:
Inclusion Criteria:

* The patient is male and has a documented diagnosis of Hunter syndrome (MPSII).
* The adult patient has completed a cognitive assessment at screening/baseline or within the previous 3 months and has been determined to have an intelligence quotient (IQ) ≥78. Note: cognitive evaluation of pediatric patients is not required.
* The adult patient or the adult patient's legally authorized representative(s) has voluntarily signed an Institutional Review Board/Independent Ethics Committee-approved informed consent form after all relevant aspects of the study have been explained and discussed.
* The pediatric patient must be scheduled to undergo a non-study related lumbar puncture or other medical or diagnostic procedure that requires the administration of general anesthesia. The pediatric patient's parent(s) or legally authorized representative(s) must have provided written informed consent (with patient assent as relevant), after all relevant aspects of the study have been explained and discussed, to allow CSF sample collection for this study in conjunction with performance of the non-study related procedure requiring general anesthesia.

Exclusion Criteria:

* The patient has a history of complications from a previous lumbar puncture(s) or technical challenges in conducting lumbar puncture.
* The patient has received a hematopoietic stem cell transplant.
* The patient has taken aspirin, non-steroidal anti-inflammatory drugs (NSAIDs), or other over-the-counter or prescription medications that could affect blood clot formation within the 7 days prior to lumbar puncture, or has ingested such medications within 7 days prior to any study-related procedure in which a change in potential blood clot formation would be deleterious.
* The patient is currently receiving treatment with intrathecal idursulfase-IT.
* The patient is currently enrolled in an interventional clinical trial.
* The patient has participated in a clinical trial of any investigational drug, including idursulfase-IT, or device within the 30 days prior to study entry.

Max Age: 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of pediatric (<18 years of age) and adult (≥18 years of age) male patients with Hunter syndrome. Up to approximately 60 patients (approximately 30 adults and 30 children) may be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-11-12 (Actual); Primary Completion 2013-12-20 (Actual); Study Completion 2013-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (7):
- United States (5):
  - Emory University, Decatur, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - University of North Carolina, Division of Genetics and Metabolism, Chapel Hill, North Carolina
  - University of Utah School of Medicine, Salt Lake City, Utah
- United Kingdom (2):
  - Central Manchester University Hospitals NHS Foundation Trust, St. Mary's Hospital, Manchester
  - Salford Royal NHS Foundation Trust, Salford

REFERENCES:
- [Background] Wraith JE, Scarpa M, Beck M, Bodamer OA, De Meirleir L, Guffon N, Meldgaard Lund A, Malm G, Van der Ploeg AT, Zeman J. Mucopolysaccharidosis type II (Hunter syndrome): a clinical review and recommendations for treatment in the era of enzyme replacement therapy. Eur J Pediatr. 2008 Mar;167(3):267-77. doi: 10.1007/s00431-007-0635-4. Epub 2007 Nov 23. PMID 18038146
- [Background] Dickson PI. Novel treatments and future perspectives: outcomes of intrathecal drug delivery. Int J Clin Pharmacol Ther. 2009;47 Suppl 1:S124-7. PMID 20040323
- [Background] Dickson P, McEntee M, Vogler C, Le S, Levy B, Peinovich M, Hanson S, Passage M, Kakkis E. Intrathecal enzyme replacement therapy: successful treatment of brain disease via the cerebrospinal fluid. Mol Genet Metab. 2007 May;91(1):61-8. doi: 10.1016/j.ymgme.2006.12.012. Epub 2007 Feb 26. PMID 17321776
- [Background] Christian J. Hendriksz, Joseph Muenzer, Barbara K. Burton, Luying Pan, Nan Wang, Hicham Naimy, Arian Pano, and Ann J. Barbier. A Cerebrospinal Fluid Collection Study in Pediatric and Adult Patients With Hunter Syndrome. Journal of Inborn Errors of Metabolism & Screening, January 2015; vol. 3

RESULTS

PARTICIPANT FLOW:
Groups:
- No Investigational Treatment or Control Group: This was an observational study for the collection and study of cerebrospinal fluid (CSF) in patients with Hunter syndrome. No investigational treatment was given.
Period: Overall Study
Arm/Group | No Investigational Treatment or Control Group
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All patients who had undergone a procedure for CSF sample collection. This included a patient who underwent unsuccessful CSF sample collection. It did not include a patient who provided a retrospective CSF sample.
Groups:
- No Investigational Treatment or Control Group: This was an observational study for the collection and study of CSF in patients with Hunter syndrome. No investigational treatment was given.
Arm/Group | No Investigational Treatment or Control Group
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants] — Age (years) at CSF sample collection
  Participants
    <=18 years | 4
    Between 18 and 65 years | 5
    >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] — Age (years) at CSF sample collection
  years | 19.36 [4.1 to 36.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
  United Kingdom | 1

OUTCOME MEASURES:

1. Primary Outcome: Levels of Total Glycosaminoglycan (GAG) in CSF
Description: The concentration of total GAG, including heparan sulfate (HS) and dermatan sulfate (DS) oligosaccharides, in CSF was measured using an enzymatic assay.
Time Frame: Day 1
Population: Pharmacodynamic Population: All patients for which an evaluable CSF sample was collected. This included a pediatric patient who was consented to provide a retrospective CSF sample.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | No Investigational Treatment or Control Group
Number analyzed (Participants) | 9
ng/mL | 816.750 [316.450 to 1317.050]

2. Secondary Outcome: Levels of GAG in Urine
Description: The levels of GAG (including sulfated DS/HS oligosaccharides) in urine were determined by the Blyscan sulfated GAG assay kit. The concentration of GAG in urine was normalized to the urine creatinine value and reported as mg GAG/mmol creatinine.
Time Frame: Day 1
Population: Pharmacodynamic Population: All patients for which an evaluable CSF sample was collected. Urinary GAG was not measured in 2 patients: 1 pediatric patient who provided a retrospective CSF sample only (no urine sample was collected) and 1 adult patient whose CSF sample was not considered evaluable and therefore their urinary GAG was not measured.
Measure: Mean (95% Confidence Interval); unit: mg GAG/mmol Creatinine
Arm/Group | No Investigational Treatment or Control Group
Number analyzed (Participants) | 8
mg GAG/mmol Creatinine | 12.458 [3.282 to 21.633]

ADVERSE EVENTS:
Groups:
- No Investigational Treatment or Control Group: This was an observational study for the collection and study of CSF in patients with Hunter syndrome. No investigational treatment was given. Safety analyses were performed in the Safety Population, which was defined as all patients who had undergone a procedure for CSF sample collection. This included a patient who underwent unsuccessful CSF sample collection; no CSF or urine GAG data were available for this adult patient.
Arm/Group | No Investigational Treatment or Control Group
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Investigational Treatment or Control Group (N=9)
Headache (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Investigational Treatment or Control Group (N=9)
Stiff Neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Pain Secondary to Surgical Procedure (Injury, poisoning and procedural complications) | 1 (1)
Difficulty Hearing in Right Ear Secondary to Neurosurgery (Injury, poisoning and procedural complications) | 1 (1)
Intermittent Headaches Post-Neurosurgery (Injury, poisoning and procedural complications) | 1 (1)
Intermittent Lower Abdomen Spasms (Gastrointestinal disorders) | 1 (1)
Intermittent Soreness Post-Surgery (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.